CLINICAL TRIAL: NCT00785135
Title: Effects of Vertical Prism on the Symptoms of Dizziness, Headache and Anxiety as Caused by Vertical Heterophoria: A Randomized, Double-blinded, Placebo-controlled, Cross-over Study
Brief Title: Effects of Prismatic Spectacle Lenses on Symptoms of Dizziness, Headache and Anxiety as Caused by Vertical Heterophoria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit - multiple reasons.- inclusion/exclusion criteria too strict was th emain reason.
Sponsor: Vision Specialists of Birmingham (Other)
Collaborators: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VSofB 20081276
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2015-12

CONDITIONS: Binocular Dysfunction; Vertical Heterophoria; Vision, Binocular; Vision Disparity
Keywords: vision, binocular; vision disparity; headache; dizziness; anxiety; neck pain; learning disorders; asthenopia; motion sickness; depth perception; gait disorder; diplopia; photophobia; agoraphobia; panic disorder
MeSH Terms: conditions — Headache; Dizziness; Anxiety Disorders; Neck Pain; Learning Disabilities; Asthenopia; Motion Sickness; Mobility Limitation; Diplopia; Photophobia; Agoraphobia; Panic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Treatment) (Active Comparator)
  Interventions: Device: Lenses containing prismatic correction
- Placebo (control) (Sham Comparator)
  Interventions: Device: Lenses not containing prismatic correction

INTERVENTIONS:
Device: Lenses containing prismatic correction — The patient will receive lenses containing prismatic correction for heterophoria, as well as correction for hyperopia, myopia and astigmatism as indicated during initial examination.
  Arms: Standard (Treatment)
Device: Lenses not containing prismatic correction — The patient will receive lenses containing correction for hyperopia, myopia and astigmatism as indicated during initial examination. The patient will not receive prismatic correction in these lenses.
  Arms: Placebo (control)

SUMMARY:
The purpose of this study is to demonstrate whether, in patients diagnosed with Vertical Heterophoria, the symptoms of dizziness, headache and / or anxiety are reduced or eliminated when a kind of correction called vertical prism is added to the patient's normal eye glass prescription.

The experiment will involve giving the patient two pairs of glasses (one pair containing the baseline prescription with vertical prism (Standard Treatment Glasses) and the other pair containing the baseline prescription but without vertical prism (Placebo Glasses)) to demonstrate which pair of glasses is most effective in reducing the symptoms of dizziness, headache and / or anxiety in these patients.

ELIGIBILITY:
Inclusion Criteria:

* First time appointment for a patient at designated optometry office for treatment of symptoms associated with Vertical Heterophoria
* Must have symptoms of dizziness or headache or both:

  * Dizziness defined as one or more of these: lightheadedness,dizziness, vertigo, feeling off-balance, lack of coordination / "clumsy", unsteadiness while walking or drifting / veering to one side while walking, motion sickness
  * Headache defined as one or more of these: pain anywhere in the head,posterior neck / upper trapezius (upper back), face, and in and / or around the eyes
* Duration of symptoms greater than 4 months
* Evaluated for these symptoms previously by at least 1 other doctor (General Practice, Family Practice, Internal Medicine, Neurology, ENT, Emergency Medicine, Pediatrics, PM&R, Ophthalmology).
* Age >14
* The patient (or their representative) must be able and willing to fill out extra paperwork
* All Patients to be seen by same Optometrist for all visits
* Must be willing to wear glasses.
* The patient (or their representative) must be able to sign informed consent
* Must have a driver for Follow Up visits where Control and Treatment Glasses are dispensed, and when Washout period is initiated
* Must have a driver for Follow Up visits where Control and Treatment Glasses are dispensed, and when Washout period is initiated
* Must have previous negative Neuroimaging (HCT or MRI) that was ordered to assess for headache and / or dizziness

Exclusion Criteria:

* Previous diagnosis of strabismus, vertical heterotropia, CN 3, 4 or 6 palsy, "lazy eye"
* Previous eye injury or eye operation (including RK and Lasik)
* Diagnosis of glaucoma
* Diagnosis of cataracts
* Diagnosis of proptosis
* Previous C-spine surgery / fusion
* Previous Rx contains prismatic correction
* >18 PD of exophoria
* > 4 PD of vertical heterophoria on Initial Exam

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evidence of change / improvement of symptoms of headache, dizziness and anxiety as demonstrated by validated, self-administered survey tools for these symptoms | Survey tools administered at baseline, 5-7 days after wearing the first pair of glasses, 5-7 days after wearing the second pair of glasses, and when treatment is completed

SECONDARY OUTCOMES:
Evidence that a new survey tool developed by the authors to assess changes / improvement in dizziness, headache and anxiety associated with Vertical Heterophoria correlates to validated, self-administered survey tools for these same symptoms | New survey tool to be administered at baseline, 5-7 days after wearing the first pair of glasses, 5-7 days after wearing the second pair of glasses, and when treatment is completed

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Rosner, MD, Principal Investigator — Vision Specialists of Birmingham
Locations (1):
- Vision Specialists of Birmingham, Birmingham, Michigan, United States